CLINICAL TRIAL: NCT05164458
Title: A Phase Ia/Ib, Open Label, Multicenter Study of the Safety and Efficacy of IBI389 Single Agent, and in Combination With Sintilimab, Administered to Patients With Advanced Malignancies
Brief Title: Safety and Efficacy of IBI389 Single Agent, and in Combination With Sintilimab, in Patients With Advanced Malignancies
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CIBI389A101
Record Dates: First submitted 2021-11-25; First posted 2021-12-20 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IBI389 (Experimental): A dose escalation stage of IBI 389 monotherapy.
  Interventions: Drug: IBI 389 Injection
- IBI 389 + sintilimab (Experimental): A dose escalation stage of IBI 389 in combination with sintilimab.
  Interventions: Drug: IBI 308 injection; Drug: IBI 389 Injection

INTERVENTIONS:
Drug: IBI 308 injection — IBI308 IV 200mg Q3W Day1
  Arms: IBI 389 + sintilimab
Drug: IBI 389 Injection — IBI 389 IV Q2~Q3W Day 1

SUMMARY:
This study is to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD) and anti-tumor activity of IBI389 as a single agent, and in combination with sintilimab, and (or) chemotherapy in patients with advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
The study consists of a dose escalation phase (Ia) and a dose expansion phase (Ib). Phase Ia is to determine the maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D) for IBI389 as a single agent, and in combination with sintilimab. Phase (Ib) is a multi-cohort trial of CLDN18.2 positive solid tumors to evaluate safety and preliminary efficacy of IBI389 in combination with sintilimab and (or) chemotherapy or IBI389 monotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Provide signed informed consent;
2. Male or female aged at 18-75 (inclusive) years;
3. Expected survival ≥12 weeks;
4. ECOG PS score 0 or 1;
5. Provide archival or fresh tissues for CLDN18.2 expression analysis;
6. Adequate laboratory parameters;
7. Suffer from advanced or metastatic malignant local solid tumors confirmed by histological diagnosis and meet the criteria of the enrolled group as follows:

Ia: The subjects for whom no standard treatment regimens are available or who is intolerable to standard treatments.

Ib: pancreatic carcinoma, gastric adenocarcinoma, advanced or metastatic solid tumors

Exclusion Criteria:

1. Participate in another interventional clinical study, except for the observational (non-interventional) clinical study or the survival follow-up phase of the interventional study.
2. Any investigational drugs received within 4 weeks prior to the first study treatment.
3. Receive the last dose of anti-tumor therapy within 4 weeks before the first dose of study therapy.
4. Immunosuppressive drugs were used within 4 weeks prior to the first administration of the study drug.
5. Medication requiring long-term systemic hormones or any other immunosuppression therapy.
6. Major surgical procedures (craniotomy, thoracotomy, or laparotomy) or unhealed wounds, ulcers, or fractures were performed within 4 weeks prior to the first dose of study therapy.
7. There was unrecovered toxicity (excluding hair loss or fatigue) according to NCI CTCAE v5.0 induced by previous antitumor therapy (24 weeks before the first dose of study), and there were unrecovered immune-related adverse events (irAE) associated with immunotherapy.
8. Primary central nervous system (CNS) malignancy, or untreated/active CNS metastases, or leptomeningeal disease.
9. History of autoimmune disease , present active autoimmune disease or inflammatory diseases
10. Present or history of pulmonary diseases such as interstitial pneumonia, pneumoconiosis, drug-related pneumonia, pulmonary fibrosis, active pulmonary infection, severely impaired pulmonary function.
11. Positive human immunodeficiency virus (HIV) test.
12. Active hepatitis B or C, or tuberculosis.
13. History of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
14. History of gastrointestinal perforation and/or fistula at 6 months prior to study inclusion.
15. Hydrothorax, ascites, and pericardial effusion with clinical symptoms requiring drainage.
16. Known history of hypersensitivity to any components of the IBI389 or Sintilimab.
17. Uncontrolled complications of disease.
18. Other acute or chronic illness, mental illness, or abnormal laboratory test values that may increase the risk of study participation or administration of study drugs, or interfere with the interpretation of study results.
19. Pregnant or nursing females.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2022-03-22 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with AEs and SAEs | up to 2 years after enrollment
  To evaluate the safety and tolerability of IBI389 alone or in combination with Sintilimab [Adverse events (AEs), Serious Adverse Events (SAEs) ]
Percentage of Participants with Dose-Limiting Toxicities (DLTs) | up to 28 Days following first dose
  To evaluate the safety and tolerability of IBI389 alone or in combination with Sintilimab.

SECONDARY OUTCOMES:
Pharmacokinetics: AUC | up to 2 years after enrollment
  The area under the curve (AUC) of serum concentration of the drug after the administration.
Cmax | up to 2 years after enrollment
  Maximum concentration (Cmax) of the drug after administration
Immunogenicity: Percentage of ADA positive subjects | up to 2 years after enrollment
  Immunogenicity: Number of Anti-Drug Antibodies (ADA) positive subjects will be counted and percentage of ADA positive subjects will be calculated to evaluate immunogenicity of IBI389.
Preliminary anti-tumor activity of IBI389 (Objective Response Rate) | up to 2 years after enrollment
  Objective Response Rate (ORR) is the percentage of Complete Response (CR) plus partial response (PR) assessed by RECIST v1.1 criteria for solid tumors.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li X, Dai R, Xu Q, Guo Z, Hu C, Sun Y, Niu Z, Hao J, Zhang M, Dai G, Hua D, Pan Y, Wang X, Wei S, Chen X, Wu Q, Zhang Y, Zhou H, Ying J, Zheng L, Bi F. Safety and preliminary efficacy results of IBI389, an anti-Claudin18.2xCD3 bispecific antibody, in patients with solid tumors and gastric or gastro-esophageal tumors: a phase 1 dose escalation and expansion study. BMC Med. 2026 Jan 16. doi: 10.1186/s12916-025-04597-8. Online ahead of print. PMID 41540424